CLINICAL TRIAL: NCT03016793
Title: Evaluation of Esthetic Satisfaction and Bone Augmentation Quality Using Purabone Added to β-tricalcium Phosphate Versus β-tricalcium Phosphate Alone in Secondry Alveolar Cleft Grafting . Randomized Controlled Clinical Trial
Brief Title: Alveolar Cleft Grafting Using Two Different Alloplastic Grafts
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamad Hamed Maklad, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pura-28568
Record Dates: First submitted 2016-12-23; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Alveolar Cleft Grafting
MeSH Terms: interventions — puerarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- puerarin and β- tricalcium phosphate (Experimental): purabone (puerarin) is an osteoinductive bone grafts used to augment bone healing.
  β- tricalcium phosphate is an osteoconductive bone graft used to augment bone healing
  Interventions: Drug: Puerarin; Drug: β- tricalcium phosphate
- β- tricalcium phosphate alone (Active Comparator): β- tricalcium phosphate is an osteoconductive bone graft used to augment bone healing
  Interventions: Drug: β- tricalcium phosphate alone

INTERVENTIONS:
Drug: Puerarin — purabone (puerarin) is a bone graft used for surgical repair of bony defects.
  Other Names: purabone
  Arms: puerarin and β- tricalcium phosphate
Drug: β- tricalcium phosphate — β- tricalcium phosphate is a bone graft used for surgical repair of bony defects
  Arms: puerarin and β- tricalcium phosphate
Drug: β- tricalcium phosphate alone — β- tricalcium phosphate is a bone graft used for surgical repair of bony defects
  Other Names: β- tricalcium phosphate
  Arms: β- tricalcium phosphate alone

SUMMARY:
P-patients with unilateral alveolar clefts I-purabone with -β-tricalcium phosphate graft C-β-tricalcium phosphate graft alone O-clinical out come Outcome name Measurement device Measurement unit Esthetic satisfaction (Primary outcome) Numerical rating scale(NRS) Number 0-10

Radiographic outcome:

Outcome name Measurment Device Measurment unite Bone volume

(Secondary out come) (CBCT)machine Cranex 3D Sordex Cubic millimeter Bone Density

(Secondary Outcome) (CBCT)machine Cranex 3D Sordex Hounsfield Unite Research Question Would purabone addition to β-tricalcium phosphate be more effective and esthetically satisfying than tricalcium phosphate alone in alveolar cleft grafting?

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral alveolar cleft indicated for bone grafting.
2. Patients age range between 8-12years.

Exclusion Criteria:

1. Patients with any systemic diseases that can affect normal bone and/or wound healing.
2. Patients with bilateral alveolar clefts.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Esthetic satisfaction | 6 months
  outcome measured by numerical scale from 1-10

SECONDARY OUTCOMES:
bone volume | 6 months
  outcome measured by cone beam computed tomography ( CBCT)
bone density | 6 months
  Outcome measured by cone beam computed tomography (CBCT)

CONTACTS AND LOCATIONS:
Overall Officials: Samar Swelam, Phd, Study Director — faculty of oral and dental medicine
Locations (1):
- Mohamad hamed Maklad, Suez, Egypt

IPD SHARING:
Plan to Share IPD: Undecided